CLINICAL TRIAL: NCT00775463
Title: DISTOL-1: Digital Ischemic Lesions in Scleroderma Treated With Oral Treprostinil Diethanolamine: A Randomized, Double-blind, Placebo-controlled, Multicenter Study
Brief Title: Digital Ischemic Lesions in Scleroderma Treated With Oral Treprostinil Diethanolamine
Acronym: DISTOL-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDE-DU-201
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: Scleroderma, Diffuse; Scleroderma, Limited; Scleroderma, Systemic; Ulcer; prostacyclin
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Limited; Ulcer | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- treprostinil diethanolamine (Experimental): Treprostinil diethanolamine sustained release tablet initiated at 0.25 mg BID and titrated up to a maximum dose of 16 mg BID or the individual's maximum tolerated dose.
  Interventions: Drug: treprostinil diethanolamine
- placebo (sugar pill) (Placebo Comparator): Matching placebo sustained release tablet initiated at 0.25 mg BID and titrated up to a maximum dose of 16 mg BID or the individual's maximum tolerated dose.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: treprostinil diethanolamine — oral sustained release tablet. Maximum tolerable dose not exceeding 16 mg twice daily (BID)
  Arms: treprostinil diethanolamine
Drug: placebo
  Arms: placebo (sugar pill)

SUMMARY:
This study will evaluate the effect of treprostinil diethanolamine (UT-15C) sustained release tablets(compared to placebo) on digital ulcers in patients with scleroderma. Treprostinil diethanolamine is an analog of prostacyclin. Prostacyclin is a naturally occuring substance produced by the cells of blood vessels that inhibits platelet aggregation, induces vasodilation, and suppresses smooth muscle proliferation. Improvement in blood flow in lower limbs and fingers would be anticipated to result in a reduction in ischemic pain, Raynaud's phenomenon and promote healing of digital ulcers and other ischemic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Subject gave voluntary written informed consent to participate in the study
* Diagnosis of systemic sclerosis (SSc) as defined by American College of Rheumatology (ACR) criteria
* Males and females age greater than 18 years at Screening
* Presence of at least one active digital ulcer (met protocol defined qualifications for active digital ulcer) at Baseline
* Females of childbearing potential willing to use a reliable form of medically acceptable contraception and have a negative pregnancy test at Screening and Baseline
* Able to communicate effectively with study personnel and willing to comply with protocol requirements

Exclusion Criteria:

* Diagnosis of pulmonary arterial hypertension (PAH)
* Body weight less than 40 kg at Screening and confirmed at Baseline
* History of postural hypotension, unexplained syncope, a blood pressure that is less than 90 mmHg systolic or 50 mmHg diastolic at Screening and Baseline
* Hemoglobin concentration less than 75% of the lower limit of the normal range at Screening
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C, or ALT greater than three times upper limit of normal
* Intractable diarrhea, or severe malabsorption, defined as greater than 15% unintentional loss of body weight in the last 6 months prior to Screening; any severe organ failure (e.g., lung, kidney), bleeding diathesis or platelet disorder, or any life-threatening condition
* Pregnant or breast-feeding
* Simultaneously fulfilled criteria for a second connective tissue disease including systemic lupus erythermatosus, rheumatoid arthritis or inflammatory myopathy
* Sympathectomy of the upper limb, involving the hand, performed within 12 months of Baseline. Sympathectomy performed on the non-target limb (hand not presenting with qualifying ulcers) or which did not include the hand, performed within 6 months of Baseline
* Receipt of prostanoid treatment (epoprostenol, treprostinil sodium, or other prostacyclin analog) within the previous 3 months of Baseline for conditions including Raynaud's phenomenon, rest pain and / or digital ulcers
* Required systemic antibiotics for infected digital ulcers within 2 weeks of Screening
* Local injection of botulinum toxin in an affected finger within 1 month prior to Baseline
* Treatment with endothelin receptor antagonists within 1 month prior to Baseline
* Patients on phosphodiasterase inhibitors, such as sildenafil or tadalafil, who have received treatment for less than 6 months prior to Baseline (unless for intermittent treatment of male erectile dysfunction)
* Treatment with statin within 1 month prior to Screening, unless for management of hyperlipidemia
* Received an investigational product within 1 month preceding Screening
* Known hypersensitivity to treprostinil diethanolamine or any of the excipients
* Tobacco or nicotine use at any level within the past 6 months prior to Screening
* Any condition or laboratory that in the opinion of the investigator might interfere with subject's participation, pose an additional risk for the subject, could prevent understanding the objectives, nature or consequences of the trial, compliance with the protocol, adherence to therapy, or that would interfere with interpretation of study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Seibold, MD, Principal Investigator — Scleroderma Research Consultants LLC, Avon, CT,
Locations (30):
- United States (24):
  - University of Alabama - Arthritis Clinical Intervention Program, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - Stanford University School of Medicine/Palo Alto VA Health Care System, Palo Alto, California
  - Denver Medical Center, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - University of Indiana School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University - Division of Rheumatology, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan Scleroderma Program, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - UMDNJ Clinical Research Center, New Brunswick, New Jersey
  - North Shore-LIJ Health System, Lake Success, New York
  - The Hospital for Special Surgery, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Dalhousie University - QEII Health Science Center, Halifax, Nova Scotia
  - St Joseph's Health Care, London, Ontario
  - McGill University, Montreal, Quebec
- United Kingdom (3):
  - Clinical Sciences Center - University Hospital, Liverpool
  - Royal Free Hospital - Center for Rheumatology, London
  - Salford Royal Hospital, Manchester

REFERENCES:
- [Derived] Mecoli CA, Perin J, Van Eyk JE, Zhu J, Fu Q, Allmon AG, Rao Y, Zeger S, Wigley FM, Hummers LK, Shah AA. Vascular biomarkers and digital ulcerations in systemic sclerosis: results from a randomized controlled trial of oral treprostinil (DISTOL-1). Clin Rheumatol. 2020 Apr;39(4):1199-1205. doi: 10.1007/s10067-019-04863-0. Epub 2019 Dec 19. PMID 31858338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited across 32 clinical trial sites in the US, Canada and UK experienced in the treatment of systemic sclerosis (SSc) and capable of conducting the trial according to ICH GCP guidance. Subjects were recruited between April 2009 and October 2010.
Groups:
- Placebo: Matching placebo sustained release tablet initiated at 0.25 mg BID and titrated up to a maximum dose of 16 mg BID or the individual's maximum tolerated dose.
Period: Overall Study
Arm/Group | Placebo | Treprostinil Diethanolamine
Started | 76 | 72
Completed | 65 | 59
Not Completed | 11 | 13
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 7 | 9
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographics and characteristics were summarized for subjects who received at least one dose of study drug. One subject in the treprostinil diethanolamine treatment group was randomized, withdrew consent and exited the study prior to taking any study medication and is not included in the summary.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treprostinil Diethanolamine | Total
Number analyzed (Participants) | 76 | 71 | 147
Age, Continuous [Mean (Full Range); unit: years] | 47.8 [20 to 74] | 49.8 [19 to 82] | 48.8 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 21 | 17 | 38
Race/Ethnicity, Customized [Number; unit: participants] — Note: A Subject can be included in more than one race category.
  participants
    Asian | 3 | 4 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 10 | 7 | 17
    White | 62 | 59 | 121
    Unknown or Not Reported | 1 | 1 | 2
SSc Classification [Number; unit: participants]
  Limited | 55 | 40 | 95
  Diffuse | 21 | 31 | 52
Years since SSc diagnosis [Mean (Full Range); unit: years] | 10.7 [0 to 30] | 10.3 [0 to 35] | 10.5 [0 to 35]

OUTCOME MEASURES:

1. Primary Outcome: Net Ulcer Burden
Description: Net ulcer burden was defined as the number of "new" or "active" digital ulcers (DU), plus the number of "indeterminate" DUs at that assessment that have previously been classified as either "active" or "new" at any earlier assessment during the study. A DU was defined as an area with visually discernable depth and a loss of continuity of epithelial coverage, which could be denuded or covered by a scab or necrotic tissue. If denuded, the DU was pronounced "active." If denudation could not be judged because of the presence of scab or necrotic tissue, DU presenting with features, including underlying pain, based on Investigator clinical judgment to be consistent with loss of epithelialization, epidermis, or dermis, and requiring treatment were designated as "active." Otherwise, the DU was pronounced "indeterminate." Only DUs distal to the proximal interphalangeal joints, volar to the equator of the finger, not localized in creases and vascular in origin were assessed.
Time Frame: Week 20
Population: The intent to treat population is all subjects that received at least one dose of study drug. Subjects were counted in the assigned group regardless of the actual treatment given. Missing values imputed by carrying last observation forward or assigning value equalling overall poorest relative change.
Measure: Median (Inter-Quartile Range); unit: ulcers
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 71
ulcers
  Baseline | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Change at Week 20 | 0.0 [-1.0 to 1.0] | -1.0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs Treprostinil Diethanolamine; A Cochran-Mantel Haenszel mean score test was used on the standardized reverse mid-ranks (overall reverse ranks divided by the number of ranks +1, or modified ridit scores; largely negative changes had ranks near 1 and largely positive changes had ranks near 0)of the residuals from an ordinary least squares regression with change in net ulcer burden at Week 20 as a linear function of Baseline PDEI or prostacyclin use (binary variable:Yes/No) and net ulcer burden at Baseline(continuous variable); Test type: Superiority or Other; p = 0.20, Cochran-Mantel-Haenszel; Hodges-Lehmann Estimate of Treatment Eff = 0.0, 95% CI 2-sided [-1.0 to 0.0]

2. Secondary Outcome: Digital Ulcer Pain VAS
Description: Digital ulcer pain was rated on a 100-mm VAS on which subjects were asked to rate their average overall hand pain during the last week. The recorded value was divided by 10, with values ranging from 0.0 (no pain) to 10.0 (unbearable pain), expressed to one decimal.
Time Frame: Week 20
Population: The intent to treat population is all subjects that received at least one dose of study drug. Subjects were counted in the assigned group regardless of the actual treatment given. Missing values imputed by carrying last observation forward or assigning value equalling overall poorest relative change. Excluded subjects without a Baseline observation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 70
units on a scale
  Baseline | 4.85 [2.75 to 6.75] | 6.00 [2.80 to 7.70]
  Change at Week 20 | -1.05 [-3.20 to 0.10] | -1.45 [-4.60 to 0.00]
Statistical Analysis 1: Comparison: Placebo vs Treprostinil Diethanolamine; The difference between treatment groups for the change from Baseline was tested using the Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney) — Analyses of secondary endpoints were descriptive in nature, no adjustments for multiplicity were made. P-values are for the purpose of describing the random imbalance between treatment groups and not to test formal hypotheses; Hodges-Lehmann Estimate of Treatment Eff = -0.40, 95% CI 2-sided [-1.40 to 0.40]

3. Secondary Outcome: Patient Global Assessment of Digital Ulcer Severity VAS
Description: Patients rated their global impression of digital ulcer severity on a 15-cm VAS from scaled 0 (no disease activity) to 100 (very severe disease).
  The term "severity" was used to measure the extent of disease activity and associated disability or discomfort the patient experienced during the indicated time period.
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 70
units on a scale
  Baseline | 57.0 [29.3 to 79.7] | 67.0 [34.7 to 78.0]
  Change at Week 20 | -24.0 [-43.0 to 0.0] | -24.3 [-63.3 to -3.3]
Statistical Analysis 1: Comparison: Placebo vs Treprostinil Diethanolamine; The VAS-global assessments were recorded in centimeters, with possible values ranging from 0.0 to 15.0. The recorded value was divided by 15, then multiplied by 100 to convert it to the VAS-Global scale, with values ranging from 0 (no disease activity) to 100 (very severe disease). The difference between treatment groups for the change from Baseline was tested using the Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Hodges-Lehmann Estimate of Treatment Eff = -9.3, 95% CI 2-sided [-21.3 to 2.7]

4. Secondary Outcome: Physician Global Assessment of Digital Ulcer Severity VAS
Description: Physicians rated their global impression of digital ulcer severity on a 15-cm VAS from scaled 0 (no disease activity) to 100 (very severe disease).
  The term "severity" was used to measure the extent of disease activity and associated disability or discomfort the patient experienced during the indicated time period.
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 70
units on a scale
  Baseline | 44.7 [26.0 to 63.3] | 47.3 [31.3 to 66.7]
  Change at Week 20 | -13.3 [-31.3 to -1.3] | -26.7 [-43.3 to -5.3]
Statistical Analysis 1: Comparison: Placebo vs Treprostinil Diethanolamine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Hodges-Lehmann Estimate of Treatment Eff = -9.3, 95% CI 2-sided [-18.0 to 0.0]

5. Secondary Outcome: Cochin Hand Function Scale (CHFS)
Description: The CHFS has been demonstrated as a reliable and valid assessment of hand function at the activity level in persons with SSc. It is comprised of 18 questions with possible integer responses of 0 (without difficulty) to 5 (impossible). The CHFS Score is simply the sum of all 18 questions, divided by the number of questions actually answered, multiplied by 18. At least 10 of the 18 questions must have been answered in order for CHFS to be calculated. Therefore, CHFS Score values can range from 0 (least limitation) to 90 (most limitation). A higher score indicates more difficulty in hand function or greater disability.
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 71
units on a scale
  Baseline | 18.5 [5.0 to 29.5] | 24.0 [11.0 to 37.0]
  Week 20 | 19.0 [4.0 to 33.5] | 21.0 [8.0 to 35.0]
Statistical Analysis 1: Comparison: Placebo vs Treprostinil Diethanolamine; The difference between treatment groups for the change from Baseline in CHFS Score were tested using the Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.47, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Hodges-Lehmann Estimate of Treatment Eff = -1.0, 95% CI 2-sided [-4.0 to 2.0]

6. Secondary Outcome: Scleroderma Health Assessment Questionnaire (SHAQ)
Description: The SHAQ is a patient self-administered instrument which has been previously validated in SSc and demonstrates meaningful clinical changes in the course of the disease over time. It is comprised of a 20 question instrument pertaining to specific activities with possible integer responses of 0 (without any difficulty) to 3 (unable to do), and five additional scleroderma-specific visual analog scale (VAS) domains (Overall Disease Activity, Raynaud's Phenomenon, Finger Ulcers, Breathing, and Intestinal Problems) with possible values ranging from 0.0 to 15.0. The 20 questions are divided into eight domains. A mean score is calculated for each domain ranging from 0 to 3. A composite HAQ DI score is calculated by dividing the summed domain scores by the number of domains answered. The composite score is reported, falling between 0 and 3 on an ordinal scale. The scores are interpreted as 0 (no impairment in function) to 3 (maximal impairment of function).
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 71
units on a scale
  Dressing & Grooming Score: Baseline (76/71) | 0.50 [0.00 to 1.00] | 1.00 [0.50 to 1.50]
  Dressing&Grooming Score:Change at Week 20 | 0.00 [0.00 to 0.00] | 0.00 [-0.50 to 0.00]
  Arising Score: Baseline (76/71) | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00]
  Arising Score: Change at Week 20 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Eating Score: Baseline (76/71) | 0.67 [0.00 to 1.00] | 0.67 [0.33 to 1.00]
  Eating Score: Change at Week 20 | 0.00 [-1.17 to 0.08] | 0.00 [-0.33 to 0.17]
  Walking Score: Baseline (76/71) | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.50]
  Walking Score: Change at Week 20 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Hygiene Score: Baseline (76/68) | 0.00 [0.00 to 0.67] | 0.33 [0.00 to 0.67]
  Hygiene Score: Change at Week 20 | 0.00 [0.00 to 0.33] | 0.00 [0.00 to 0.33]
  Reach Score: Baseline (76/68) | 0.00 [0.00 to 1.00] | 0.50 [0.00 to 1.00]
  Reach Score: Change at Week 20 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Grip Score: Baseline (76/68) | 0.33 [0.00 to 0.67] | 0.33 [0.17 to 1.00]
  Grip Score: Change at Week 20 | 0.00 [0.00 to 0.33] | 0.00 [-0.33 to 0.00]
  Activity Score: Baseline (76/68) | 0.33 [0.00 to 1.00] | 0.67 [0.00 to 1.00]
  Activity Score: Change at Week 20 | 0.00 [0.00 to 0.33] | 0.00 [0.00 to 0.17]
  HAQ Aggregate Score: Baseline (76/68) | 0.34 [0.10 to 0.77] | 0.53 [0.26 to 0.81]
  HAQ Aggregate Score: Change at Week 20 | 0.00 [-0.07 to 0.13] | -0.03 [-0.16 to 0.12]
  Hand Function Aggregate Score: Baseline (76/68) | 0.39 [0.11 to 0.69] | 0.56 [0.28 to 0.86]
  Hand Function Aggregate Score: Change at Week 20 | 0.00 [-0.06 to 0.17] | 0.00 [-0.22 to 0.11]
  Raynaud's Phenomenon VAS Score: Baseline (75/71) | 0.12 [0.00 to 0.64] | 0.18 [0.02 to 0.80]
  Raynaud's Phenomenon VAS Score: Change at Week 20 | 0.00 [-0.14 to 0.08] | 0.00 [-0.14 to 0.14]
  Intestinal Problems VAS Score: Baseline (75/70) | 0.20 [0.00 to 0.70] | 0.11 [0.02 to 0.62]
  Intestinal Problems VAS Score: Change at Week 20 | 0.00 [-0.10 to 0.24] | 0.11 [-0.02 to 0.72]
  Digital Ulcer VAS Score: Baseline (76/71) | 1.43 [0.49 to 2.09] | 1.50 [0.68 to 2.28]
  Digital Ulcer VAS Score: Change at Week 20 | -0.34 [-0.92 to 0.00] | -0.56 [-1.36 to 0.00]
  Breathing Problems VAS Score: Baseline (76/71) | 1.54 [0.95 to 2.31] | 2.16 [0.96 to 2.54]
  Breathing Problems VAS Score: Change at Week 20 | -0.50 [-1.15 to 0.00] | -0.84 [-2.14 to -0.20]
  Pain VAS Score: Baseline (76/69) | 1.27 [0.57 to 1.91] | 1.54 [0.54 to 2.16]
  Pain VAS Score: Change at Week 20 | -0.26 [-0.93 to 0.11] | -0.34 [-1.44 to 0.00]
  Overall Disease VAS Score: Baseline (76/71) | 1.22 [0.67 to 1.87] | 1.52 [0.74 to 2.12]
  Overall Disease VAS Score: Change at Week 20 | -0.18 [-0.60 to 0.04] | -0.32 [-1.00 to 0.10]

7. Secondary Outcome: Modified Rodnan Skin Score (mRSS)
Description: The skin thickening was assessed by the Investigator in 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Each area was scored 0-3; 0 representing normal skin and 3 being severe thickening. The mRSS was the sum of the individual skin assessment scores: possible range of 0-51; 0 (no thickening) to 51 (severe thickening in all 17 areas) .
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 71
units on a scale
  Baseline | 6.0 [3.0 to 12.0] | 8.0 [5.0 to 14.0]
  Week 20 | 6.0 [3.0 to 12.0] | 6.0 [3.0 to 15.0]
Statistical Analysis 1: Comparison: Placebo vs Treprostinil Diethanolamine; he difference between treatment groups for the change from Baseline and at Week 20 in the mRSS was tested using the Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney); Hodges-Lehmann Estimate of Treatment Eff = 0.0, 95% CI 2-sided [0.0 to 1.0]

8. Secondary Outcome: Short-Form McGill Pain Questionnaire
Description: The SF-MPQ assessment has three component scores: the pain rating index (PRI), a pain visual analogue numerical scale (Pain VAS) and the present pain intensity (PPI). PRI is calculated by summing the responses (0=None to 3=Severe) to the 15 questions describing pain during the previous week and rated on an intensity scale as 0= none, 1= mild, 2= moderate or 3= severe and has possible values ranging from 0 to 45. The Pain VAS is a 100 mm VAS on which subjects were asked to rate pain during the previous week with values ranging from no pain (0.0) to worst possible pain (10.0). The PPI rated pain on a 6-point category scale from 0 (no pain) to 5 (excruciating pain).
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 74 | 68
units on a scale
  Total Pain Rating Index Score Change at Week 20 | -4.0 [-8.0 to 1.0] | -3.0 [-12.0 to 0.0]
  Pain VAS Score Change at Week 20 | -0.6 [-2.9 to 0.3] | -1.1 [-4.4 to 0.2]
  Present Pain Intensity Score Change at Week 20 | 0.0 [-1.0 to 0.0] | -1.0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs Treprostinil Diethanolamine; P value for Total Pain Rating Index Score; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney) — P value for Total Pain Rating Index Score; Hodges-Lehmann Estimate of Treatment Eff = -1.0, 95% CI 2-sided [-3.0 to 2.0]
Statistical Analysis 2: Comparison: Placebo vs Treprostinil Diethanolamine; P value for Pain VAS; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney) — P value for Pain VAS; Hodges-Lehmann Estimate of Treatment Ef = -0.6, 95% CI 2-sided [-1.6 to 0.3]
Statistical Analysis 3: Comparison: Placebo vs Treprostinil Diethanolamine; P value for Total Pain Rating Index Score; Test type: Superiority or Other; p = 0.10, Wilcoxon (Mann-Whitney) — P value for Total Pain Rating Index Score; Hodges-Lehmann Estimate of Treatment Eff = 0.0, 95% CI 2-sided [-1.0 to 0.0]

9. Secondary Outcome: Patient Impression of Change (PIC) Questionnaire
Description: The PIC questionnaire consisted of three Likert items that asked the subject to rate changes in their digital ulcer, Raynaud's phenomenon and disease status since their last visit on a seven-level scale (very much improved, much improved, somewhat improved, same, somewhat worse, much worse and very much worse).
Time Frame: Week 20
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Placebo- Digital Ulcer Response; Placebo- Raynaud's Phenomenon Response; Placebo- Overall Disease Status Response: Matching placebo sustained release tablet initiated at 0.25 mg BID and titrated up to a maximum dose of 16 mg BID or the individual's maximum tolerated dose.
- Treprostinil Diethanolamine- Digital Ulcer Response; Treprostinil Diethanolamine- Raynaud's Phenomenon Response; Treprostinil Diethanolamine- Overall Disease Status Response: Treprostinil diethanolamine sustained release tablet initiated at 0.25 mg BID and titrated up to a maximum dose of 16 mg BID or the individual's maximum tolerated dose.
Arm/Group | Placebo- Digital Ulcer Response | Treprostinil Diethanolamine- Digital Ulcer Response | Placebo- Raynaud's Phenomenon Response | Treprostinil Diethanolamine- Raynaud's Phenomenon Response | Placebo- Overall Disease Status Response | Treprostinil Diethanolamine- Overall Disease Status Response
Number analyzed (Participants) | 76 | 71 | 76 | 71 | 76 | 71
participants
  Very Much Improved | 5 | 9 | 0 | 3 | 0 | 3
  Much Improved | 11 | 15 | 4 | 12 | 5 | 17
  Somewhat Improved | 20 | 14 | 12 | 20 | 22 | 13
  Same | 24 | 21 | 40 | 30 | 30 | 27
  Somewhat Worse | 14 | 8 | 17 | 4 | 18 | 10
  Much Worse | 1 | 3 | 1 | 1 | 0 | 0
  Very Much Worse | 1 | 1 | 2 | 1 | 1 | 1

10. Secondary Outcome: Short Form 36
Description: Change in patient quality of life was measured by the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36), a self-administered questionnaire covering eight areas: physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health. For each area, the score range from 0 (poorer health status) to 100 (better health status). The SF-36 is one of the most widely used and validated instruments to assess quality of life in patients with systemic illnesses. A decrease (negative change) in a domain score corresponds to deterioration.
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 71
units on a scale
  Physical Component: Baseline | 55.0 [39.5 to 67.5] | 50.7 [35.1 to 62.9]
  Physical Component: Change at Week 20 | 2.8 [-5.3 to 10.9] | 3.8 [-2.1 to 10.3]
  Physical Functioning: Baseline | 62.5 [30.0 to 80.0] | 60.0 [35.0 to 75.0]
  Physical Functioning: Change at Week 20 | 0.0 [-5.0 to 10.0] | 0.0 [-10.0 to 10.0]
  Role-Physical: Baseline | 54.4 [37.5 to 72.5] | 50.0 [25.0 to 70.0]
  Role-Physical: Change at Week 20 | 0.0 [-10.0 to 17.5] | 0.0 [0.0 to 22.5]
  Bodily Pain: Baseline | 57.5 [33.8 to 67.5] | 45.0 [32.5 to 75.0]
  Bodily Pain: Change at Week 20 | 10.0 [-5.0 to 21.3] | 10.0 [-2.5 to 22.5]
  General Health: Baseline | 42.0 [34.0 to 65.0] | 45.0 [30.0 to 63.0]
  General Health: Change at Week 20 | 0.0 [-9.5 to 5.0] | 0.0 [-5.0 to 6.0]
  Mental Component: Baseline | 68.3 [54.1 to 77.4] | 64.2 [49.2 to 76.1]
  Mental Component: Change at Week 20 | 2.6 [-8.6 to 11.0] | 4.0 [-4.0 to 15.7]
  Vitality: Baseline (75/71) | 50.0 [31.3 to 62.5] | 43.8 [25.0 to 61.3]
  Vitality: Change at Week 20 | 0.0 [-6.3 to 7.5] | 1.3 [-6.3 to 17.5]
  Social Functioning: Baseline | 72.5 [50.0 to 87.5] | 62.5 [50.0 to 85.0]
  Social Functioning: Change at Week 20 | 0.0 [-12.5 to 13.8] | 10.0 [0.0 to 22.5]
  Role-Emotional: Baseline | 70.0 [60.8 to 95.0] | 80.0 [50.0 to 100.0]
  Role-Emotional: Change at Week 20 | 0.0 [-5.8 to 11.7] | 0.0 [-1.7 to 13.3]
  Mental Health: Baseline (75/71) | 69.0 [52.0 to 84.0] | 64.0 [54.0 to 79.0]
  Mental Health: Change at Week 20 | 2.0 [-6.0 to 11.0] | 3.0 [-5.0 to 16.0]

11. Secondary Outcome: Time to Ulcer Healing- Percentage of Subjects With Complete Healing
Description: A subject was counted as having all ulcers completely healed at the earliest assessment for which all ulcers are designated as "healed" and no new ulcers appeared for the remainder of the trial.
Time Frame: Week 20
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 71
percentage of participants
  Cardinal Ulcer Healed | 61 | 62
  All Ulcers Healed | 41 | 49

12. Secondary Outcome: Time to Ulcer Healing
Description: A subject was counted as having all ulcers completely healed at the earliest assessment for which all ulcers are designated as "healed" and no new ulcers appeared for the remainder of the trial. The time to complete healing of all ulcers were calculated as the number of days from randomization to the date of these respective assessments, provided that complete healing was achieved during the study.
Time Frame: Week 20
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Treprostinil Diethanolamine
Number analyzed (Participants) | 76 | 71
days
  Time to Cardinal Ulcer Healing | 83.2 (37.9) | 76.3 (35)
  Time to All Ulcers Healed | 96.7 (39.7) | 90.2 (35.6)

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Placebo | Treprostinil Diethanolamine
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/71
Serious Adverse Events (participants affected / at risk) | 4/76 | 9/71
Other Adverse Events (participants affected / at risk) | 74/76 | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Treprostinil Diethanolamine (N=71)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Treprostinil Diethanolamine (N=71)
Headache (Nervous system disorders) | 32 (46) | 52 (71)
Diarrhoea (Gastrointestinal disorders) | 16 (21) | 40 (48)
Fatigue (General disorders) | 15 (15) | 16 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (16) | 12 (13)
Infected skin ulcer (Skin and subcutaneous tissue disorders) | 10 (13) | 13 (16)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4 (5) | 17 (20)
Flushing (Vascular disorders) | 3 (3) | 17 (19)
Oedema peripheral (General disorders) | 11 (12) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (11)
Vomiting (Gastrointestinal disorders) | 4 (5) | 12 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 11 (13)
Dizziness (Nervous system disorders) | 8 (9) | 8 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (9)
Pain (General disorders) | 1 (1) | 12 (18)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 10 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 4 (4)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (7) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (6)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3)
Localised infection (Infections and infestations) | 5 (5) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 5 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 5 (5)
Urinary tract infection (Renal and urinary disorders) | 4 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (3)
Migraine (Nervous system disorders) | 2 (2) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (5)
Paraesthesia (Nervous system disorders) | 1 (1) | 5 (6)
Chest pain (General disorders) | 4 (4) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (16) | 42 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other